CLINICAL TRIAL: NCT04060966
Title: Neural Mechanisms of Cost and Benefit Integration During Decision-Making, Aim 2: Acute & Lifetime Stress
Status: Completed | Type: Observational
Sponsor: NYU Langone Health (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Other Study IDs: 18-01945; 7R01DA038063-06 (NIH)
Record Dates: First submitted 2019-08-16; First posted 2019-08-19 (Actual); Last update posted 2023-07-25 (Actual); Status verified 2023-07

CONDITIONS: Healthy
MeSH Terms: interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Cohort 1: Stress Task: Participants in Cohort 1 randomized to the stress task will complete the Cold-Pressor Task (CPT), which requires the continuous submersion of the forearm in ice-water (0-4°C) for 3 minutes in the presence of an experimenter. After the CPT, participants will complete a decision-making task. During the decision-making task, participants will do one of the following: evaluate different features of foods/monetary prizes in 'rating trials', choose between pairs or bundles of snack foods in 'choice trials', bid for the chance to win foods/monetary prizes or bid to remove certain foods from their choice menu in 'auction trials', or choose between pairs of monetary lotteries in 'lottery trials'.
  Interventions: Behavioral: Cold-Pressor Task (CPT)
- Cohort 1: Control: Participants in Cohort 1 randomized to the Control group will complete a matching control task to the CPT, which involves continuous submersion of the forearm in warm water, ~30°C, for 3 minutes. After the control CPT, participants will complete a decision-making task. During the decision-making task, participants will do one of the following: evaluate different features of foods/monetary prizes in 'rating trials', choose between pairs or bundles of snack foods in 'choice trials', bid for the chance to win foods/monetary prizes or bid to remove certain foods from their choice menu in 'auction trials', or choose between pairs of monetary lotteries in 'lottery trials'.
  Interventions: Behavioral: Control CPT
- Cohort 2: Stress Task + fMRI: Participants in Cohort 2 randomized to the Stress task will complete the CPT, which requires the continuous submersion of the forearm in ice-water (0-4°C) for 3 minutes in the presence of an experimenter. After the CPT, participants will complete decision-making tasks while being scanned via functional MRI (fMRI). The tasks will involve attending to auditory and/or visual stimuli on a computer. On each trial, different food items and different amounts of time (1-60 minutes) will be presented and participants will be asked to indicate how much they would pay from their $10 study endowment to avoid spending the trial's stated amount of time with the snack food.
  Interventions: Behavioral: Cold-Pressor Task (CPT); Device: fMRI
- Cohort 2: Control + fMRI: Participants in Cohort 2 randomized to the Control group will complete a matching control task to the CPT, which involves continuous submersion of the forearm in warm water, ~30°C, for 3 minutes. After the control CPT, participants will complete decision-making tasks while being scanned via functional MRI (fMRI). The tasks will involve attending to auditory and/or visual stimuli on a computer. On each trial, different food items and different amounts of time (1-60 minutes) will be presented and participants will be asked to indicate how much they would pay from their $10 study endowment to avoid spending the trial's stated amount of time with the snack food.
  Interventions: Behavioral: Control CPT; Device: fMRI
- Cohort 3: M-Turk Survey: Participants in Cohort 3 will access the Amazon Mechanical Turk (M-Turk) platform, where they can search for available surveys ('HITs') to complete for payment on the M-Turk website. After completing the surveys, participants will complete the Stress and Adversity Inventory (STRAIN) questionnaire.

INTERVENTIONS:
Behavioral: Cold-Pressor Task (CPT) — The CPT involves participants submerging their dominant forearm in ice-water (0-4°C) for 3 minutes.
  Groups: Cohort 1: Stress Task; Cohort 2: Stress Task + fMRI
Behavioral: Control CPT — The control CPT involves participants submerging their dominant forearm in warm water (~30°C) for 3 minutes.
  Groups: Cohort 1: Control; Cohort 2: Control + fMRI
Device: fMRI — Participants in the neuroimaging cohort will complete up to two fMRI experimental sessions on different days, with at least a day between sessions, each lasting approximately 2 hours. Imaging data will be collected with a Prisma 3T head- only scanner equipped with a head coil from Nova Medical.
  Groups: Cohort 2: Control + fMRI; Cohort 2: Stress Task + fMRI

SUMMARY:
The central aim of this study is to characterize how the costs of acute and lifetime stress affect the neural architecture for decision-making in healthy humans. Investigators will use behavioral choice paradigms to measure how the costs of stress influence decisions about rewards (e.g., foods, money) as well as decisions about the use of self-control strategies. They will further examine associations between these stress measures and other decision variables commonly studied in our lab which have well-understood mechanisms, such as risk preferences. This behavioral work lays the foundation for an fMRI experiment that combines our measures of the behavioral costs of stress with neural measures of brain changes. Acute stress will be measured using a physiological stressor (cold-pressor task) coupled with saliva sample collection for cortisol analysis. Lifetime stress will be measured using a computerized life stress survey. We will study three cohorts: One purely behavioral cohort will be examined on-site (n=60). In a smaller subset of participants (n=40), investigators will measure neural activity changes in relevant brain areas as measured with MRI during decisions to use self-control in the presence of rewards. In a larger sample (n=500) the correlation between participants' risk preferences and lifetime stress exposure at scale using Amazon Mechanical Turk subjects will be measured.

ELIGIBILITY:
Inclusion Criteria:

* English as a native language
* Corrected-to-normal vision
* Individuals on diets to maintain or lose weight, or those not on a diet
* All races, ethnicities, and cultures

Exclusion Criteria:

* For all fMRI studies we will exclude participants who meet one of the standard CBI MRI exclusion criteria (see attached exclusion questionnaire) prior to participation. This screening questionnaire will be administered prior to scheduling the study, and once again before the scanner session during the second consenting procedure.
* History of and/or medication for neurological or psychiatric disorders
* High blood pressure, heart condition or related medical conditions
* Diabetes, metabolic disorders, history of eating disorders, or food allergies
* Pregnancy
* Handedness (this has been shown be indicative of variations in brain circuitry)
* Since we will measure stress hormones, subjects currently taking corticosteroids or beta-blockers will be ineligible to participate, as these medications have been found to dramatically alter stress hormone levels.
* Furthermore, evidence suggests that fluctuations in bodily hormones (such as that induced through hormonal contraceptives or different stages of menstrual cycle phase) can affect stress hormone levels (Tersman, Collins, & Eneroth, 1991; Kirschbaum et al, 1999; Andreano, Arjomanid, Cahill, 2008). In order to account for hormonal differences, we will ask female participants if they are taking oral contraceptives. Likewise, we propose to use a simple, non-invasive questionnaire to determine cycle phase, as in McCormick & Teillon, 2001. We may need to exclude on the basis of whether or not female participants use hormone-based contraceptives, which, for the reason stated above, could be a potential confound.
* In some cases, we will pre-screen subjects to ensure they are on a diet to maintain or lose weight in order to examine how dietary and health goals influence decisions about self-control and rewards.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Participants will be healthy males and females between ages of 18-64 reflecting the demographics of NYU Washington Square and New York area.
Sampling Method: Non-Probability Sample
Enrollment: 397 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2022-08-01 (Actual); Study Completion 2022-08-01 (Actual)

PRIMARY OUTCOMES:
Amount in Dollars ($) Participants are Willing to Allocate to Avoid Use of Self-Control during Decision-Making Task | Up to 2 Hours
  Amount participants would be willing to spend to avoid use of self-control will be evaluated during a decision-making task in Cohorts 1 and 2.
Stress and Adversity Inventory (STRAIN) Overall Severity Score | 60 Minutes
  Cumulative lifetime stress will be quantified as a score (Overall Severity Score; OSS) derived from the Stress and Adversity Inventory (STRAIN) questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Paul Glimcher, PhD, Principal Investigator — New York Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States

DOCUMENTS (1):
  • Informed Consent Form (2019-04-22): https://cdn.clinicaltrials.gov/large-docs/66/NCT04060966/ICF_000.pdf